CLINICAL TRIAL: NCT04439682
Title: The Effects of Exercise on Some Biochemical Parameters in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Research Assistant, Firat University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97132852/050.01.04/
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Biochemical Parameters; exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Aerobic exercise will be performed for a single session
  Interventions: Other: Aerobic exercise
- Control group (Active Comparator): Aerobic exercise will be performed to healthy population for a single session
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise will be performed to all participants for a single session. Maximum heart rate was calculated for each subject (220 - age) and a heart rate monitor (Polar FT 100, China) will be used to follow subjects' heart rate during aerobic exercise.

SUMMARY:
Background: RA may progress with articular and non-articular involvement.Depression prevelance is found to increase for RA patients according to healthy population and to be correlated with pain, decreased quality of life, fatigue and physical disability.BDNF level was found significantly lower in RA patients with depression. Aim of this study is to investigate the variation of BDNF, VEGF, TNF- α, IL-6, IL-1β, irisin and α- Klotho levels following acute exercise.

Methods: This study included 45 RA patients and 45 age and sex matched healthy controls. Blood samples from all subjects were taken and centrifuged before and immediately after the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged between 18-65 years,
* Patients who got diagnosed according to American College of Rheumatology criteria
* Patients who were being followed at Firat University Department of Rheumatology

Exclusion Criteria:

* Patients who had regular exercise habits, malignancy, pregnancy, incorporation,
* Patients who took anti-TNF treatment
* Patients who had changes of medical treatment in last 3 months
* Patients who diagnosed with Fibromyalgia Syndrome and Osteoarthritis for lower extremity
* Patients who had cardiac symptoms according to New York Heart Association
* Patients who had dysfunction that can prevent physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-17 (Estimated); Primary Completion 2020-09-17 (Estimated); Study Completion 2021-06-17 (Estimated)

PRIMARY OUTCOMES:
Irisin | 1 minute
  Blood samples from all subjects will be taken and centrifuged before and immediately after the exercise intervention. Obtained serums will be stored at the laboratories of Firat University.

SECONDARY OUTCOMES:
BDNF, VEGF, TNF- α, IL-6, IL-1β and α- Klotho | 1 minute
  Blood samples from all subjects will be taken and centrifuged before and immediately after the exercise intervention. Obtained serums will be stored at the laboratories of Firat University.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimsholm O, Rantapaa-Dahlqvist S, Dalen T, Forsgren S. BDNF in RA: downregulated in plasma following anti-TNF treatment but no correlation with inflammatory parameters. Clin Rheumatol. 2008 Oct;27(10):1289-97. doi: 10.1007/s10067-008-0910-4. Epub 2008 May 17. PMID 18484150
- [Background] Szuhany KL, Bugatti M, Otto MW. A meta-analytic review of the effects of exercise on brain-derived neurotrophic factor. J Psychiatr Res. 2015 Jan;60:56-64. doi: 10.1016/j.jpsychires.2014.10.003. Epub 2014 Oct 12. PMID 25455510
- [Derived] Ercan Z, Deniz G, Yentur SB, Arikan FB, Karatas A, Alkan G, Koca SS. Effects of acute aerobic exercise on cytokines, klotho, irisin, and vascular endothelial growth factor responses in rheumatoid arthritis patients. Ir J Med Sci. 2023 Feb;192(1):491-497. doi: 10.1007/s11845-022-02970-7. Epub 2022 Mar 16. PMID 35296975